CLINICAL TRIAL: NCT07166172
Title: North American Fetal Therapy Network Prospective Registry for Long-term Outcome Following Fetoscopic Endoluminal Tracheal Occlusion in Severe Left and Right Congenital Diaphragmatic Hernia
Brief Title: Prospective Registry for Long-term Outcomes Following FETO in Severe Left and Right CDH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00495298
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Congenital Diaphragmatic Hernia; Congenital Abnormalities; Neonatal Diseases and Abnormalities; Hernia, DIaphragmatic, Congenital; Internal Hernia; Hernia; Pathological Conditions, Anatomical; Pathological Conditions, Signs and Symptoms
Keywords: Fetoscopic Endoluminal Tracheal Occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Congenital Abnormalities; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hernia, Diaphragmatic; Internal Hernia; Hernia; Pathological Conditions, Anatomical; Pathological Conditions, Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fetal Treatment Arm (FETO Group) (Experimental)
  Interventions: Device: Fetal Treatment Arm (FETO Group)
- Expectant Management Arm (Control Group) (No Intervention): Standard of care treatment for babies with congenital diaphragmatic hernia.

INTERVENTIONS:
Device: Fetal Treatment Arm (FETO Group) — Participants will undergo FETO surgery between 27 weeks 0 days to 29 weeks 6 days gestation. The FETO intervention involves two procedures: (1) inserting a balloon into the fetal trachea, and (2) removing the balloon before delivery. After the first FETO procedure, participants will be monitored weekly by ultrasound. Removal of the balloon will be performed at 34 weeks 0 days to 34 weeks 6 days. Planned delivery will occur after 37 weeks. The follow-up phase will be conducted from birth to 24 months of age.
  Other Names: Fetal Endoluminal Tracheal Occlusion (FETO)
  Arms: Fetal Treatment Arm (FETO Group)

SUMMARY:
The purpose of this study is to evaluate successful placement and removal of Fetoscopic Endoluminal Tracheal Occlusion (FETO) device in cases of intrathoracic liver herniation with isolated left congenital diaphragmatic hernia (LCDH) with Observed/Expected (O/E) Lung to Head Circumference Ratio (LHR) < 30% or isolated right congenital diaphragmatic hernia (RCDH) with O/E LHR < 45%,to compare survival to discharge from the neonatal intensive care units (NICU), between fetuses with intrathoracic liver herniation and isolated LCDH with O/E LHR < 30% that receive FETO procedure performed at 27 weeks 0 days to 29weeks 6 days of gestation to those with intrathoracic liver herniation, isolated LCDH and o/e LRH < 30% that undergo expectant management, to compare the neonatal survival rate to discharge from the neonatal intensive care units (NICU), between fetuses with intrathoracic liver herniation, isolated RCHD with o/e LHR < 45% that undergo FETO procedure performed at 27 weeks 0 days to 29 weeks 6 days gestation to those with intrathoracic liver herniation, isolated RCHD and o/e LHR < 45% that elect to proceed with expectant management, to evaluate the frequency of maternal and fetal complications associated with FETO procedure, to evaluate whether the FETO procedure is associated with reduced long-term mortality and morbidities in isolated LCDH survivors with o/e LHR <30% when compared to isolated LCDH with o/e LRH <30% that undergo expectant management where all fetuses were found to have intrathoracic liver herniation and to evaluate whether the FETO procedure is associated with reduced long-term mortality and morbidities in isolated RCDH survivors with o/e LHR ≤ 45% when compared to isolated RCHD with LHR < 45% that undergo expectant management where all fetuses were found to have intrathoracic liver herniation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are able to consent
* Singleton pregnancy
* Normal Karyotype, chromosomal microanalysis (CMA) with non-pathologic variants, whole exome sequencing (WES) or whole genome sequencing (WGS) . Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Gestational age at enrollment is prior to 296 wks.
* Intrathoracic liver herniation
* Isolated left CDH with o/e LHR < 30% at enrollment (180 to 295 wks.) or
* Isolated RCDH with o/e LHR < 45% at enrollment (180 to 295 wks.)
* Cervical length by transvaginal ultrasound > 20 mm within 24 hours prior to FETO procedure
* Patient meets psychosocial criteria
* Informed consent understood

Exclusion Criteria:

* History of natural rubber latex allergy
* Preterm labor, cervix shortened (<20 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa.
* Psychosocial ineligibility, precluding consent:

  1. Inability to reside within 30 minutes of Johns Hopkins Hospital Center for Fetal Therapy.
  2. The patient does not have a support person (e.g., spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at Johns Hopkins Hospital Center for Fetal Therapy.
* Bilateral CDH, isolated left sided CDH with O/E LHR ≥ 30% (measured at 180 to 295 weeks), isolated right sided CDH with O/E LHR > 45% (measured at 180 to 295 weeks), as determined by ultrasound
* No liver herniation into thoracic cavity
* Additional fetal anomaly and chromosomal abnormalities by ultrasound, MRI, or echocardiogram at the fetal treatment center. Exclude chromosomal abnormalities, associated anomalies recognized to alter survival prognosis (i.e., CDH and congenital heart disease) or presence of an underlying genetic syndrome (i.e., Fryns).
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Uterine anomalies such as large or multiple fibroids or Mullerian duct abnormality
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality. or participation in this trial in a previous pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of successful placement of FETO device | 10-60 minutes after surgery begins
Number of successful removal of FETO device | Immediately after the procedure (about 1 hour after start of surgery)
Number of FETO procedure complications | End of study (24 months)
  Complications include: Failure FETO insertion procedure, FETO device dislodgement potentially requiring a second FETO insertion, Fetal intraoperative injury, Procedural hemorrhage, Bleeding from insertion site or Abruptions, Post-procedural hemorrhage PPROM, Preterm delivery, Chorioamnion separation, Chorioamnionitis, Polyhydramnios, Oligohydramnios, Emergent removal due to obstetrical complication, Failed percutaneous or fetoscopic removal requiring cesarean section or exit procedure for removal, Neonatal death due to asphyxia if delivery before FETO removal, and Non-reassuring fetal heart rate monitoring.
Number of neonates that survived | From delivery to hospital discharge
  Neonatal survival to discharge

SECONDARY OUTCOMES:
Number of infants that survived | 6 months
Number of infants that survived | 12 months
Number of infants that survived | 18 months
Number of infants that survived | 24 months
Number of infants that show presence of pulmonary hypertension | 6 months
Number of infants that show presence of pulmonary hypertension | 12 months
Number of infants that show presence of pulmonary hypertension | 18 months
Number of infants that show presence of pulmonary hypertension | 24 months
Number of infants that show need for supplemental oxygen | 6 months
Number of infants that show need for supplemental oxygen | 12 months
Number of infants that show need for supplemental oxygen | 18 months
Number of infants that show need for supplemental oxygen | 24 months
Number of infants that show periventricular leukomalacia | At less than 2 months postnatally
Number of Infants that develop sepsis | 6 months
Number of Infants that develop sepsis | 12 months
Number of Infants that develop sepsis | 18 months
Number of Infants that develop sepsis | 24 months
Number of infants that develop Intraventricular hemorrhage (grade 0-III) | 6 months
Number of infants that develop Intraventricular hemorrhage (grade 0-III) | 12 months
Number of infants that develop Intraventricular hemorrhage (grade 0-III) | 18 months
Number of infants that develop Intraventricular hemorrhage (grade 0-III) | 24 months
Number of infants that develop retinopathy of prematurity (grade 3 or higher) | 6 months
Number of infants that develop retinopathy of prematurity (grade 3 or higher) | 12 months
Number of infants that develop retinopathy of prematurity (grade 3 or higher) | 18 months
Number of infants that develop retinopathy of prematurity (grade 3 or higher) | 24 months
Number of infants that develop gastro-esophageal reflux | 6 months
Number of infants that develop gastro-esophageal reflux | 12 months
Number of infants that develop gastro-esophageal reflux | 18 months
Number of infants that develop gastro-esophageal reflux | 24 months
Number of infant hospital readmissions | End of study (24 months)
Cause of infant hospital readmissions | End of study (24 months)
Number of infants that show childhood growth failure | 6 months
Number of infants that show childhood growth failure | 12 months
Number of infants that show childhood growth failure | 18 months
Number of infants that show childhood growth failure | 24 months
Number of infants that show recurrence of CDH repair | 6 months
Number of infants that show recurrence of CDH repair | 12 months
Number of infants that show recurrence of CDH repair | 18 months
Number of infants that show recurrence of CDH repair | 24 months
Number of infants that develop bowel obstruction | 6 months
Number of infants that develop bowel obstruction | 12 months
Number of infants that develop bowel obstruction | 18 months
Number of infants that develop bowel obstruction | 24 months
Number of infants that show neurodevelopmental delay as assessed by the Bayley Scales of Infant and Toddler Development-III(BSID) | 24 months
  Three domains will be measured as follows: Cognitive Scale, Language Scale (Receptive and Expressive) and Motor Scale (Fine and Gross Motor Skills). Scores are derived by converting raw scores from completed tasks into scale scores and composite scores. These scores are then utilized to assess the child's performance in relation to norms established based on typically developing children of the same age
  Mean score of 100 (SD=15) at the 50th percentile signifies mid-average functioning.
  Scores below 85 (1 SD below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay.
  Score below 70 (2 SD below the mean), at the second percentile, indicate moderate to severe impairment.
  In general, scores falling in the lowest 10th percentile indicate developmental delay
Number of infants that develop bronchopulmonary dysplasia | 6 months
Number of infants that develop bronchopulmonary dysplasia | 12 months
Number of infants that develop bronchopulmonary dysplasia | 18 months
Number of infants that develop bronchopulmonary dysplasia | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Baschat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No